CLINICAL TRIAL: NCT01639534
Title: Biomarkers of Ischemia: Xanthine, Hypoxanthine and Inosine Levels During Carotid Stenting Procedures
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: HM12941
Record Dates: First submitted 2012-07-10; First posted 2012-07-12 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Identify the Presence of a Marker of Ischemia/Hypoperfusion of the Brain Via Peripheral Blood; Ischemia/Hypoperfusion of Brain
Keywords: Biomarkers of ischemia; Carotid Stenting procedure; Levels Xanthine Hypoxanthine and Inosine; peripheral blood
MeSH Terms: conditions — Ischemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — An aliquot of each sample will be stored for potentialconfirmatory reanalysis in the future at this or a contracted insitution.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Biomarkers, Carotid Stenting, Blood sample: Subjects requiring Carotid Stenting Procedure at Virginia Commonwealth University/Medical College of Virginia Health Systems

SUMMARY:
The purpose of the study is to determine if a new blood test can help the doctor determine if there is brain injury or ischemia. Ischemia occurs when not enough oxygen gets to the brain. In this study the investigators are analyzing your blood for a new test that might help doctors decide if symptoms are from a neurologic problem.

DETAILED DESCRIPTION:
We will compare a new blood test with routine tests that the doctor will order as part of your normal care. This study will measure new biomarkers (biomarker is a specific distinguishing feature used to measure or indicate the effects or progress of a disease or condition) of neurologic stress called xanthine, hypoxanthine, and inosine. Blood will be drawn as a part of the study to measure these biomarker levels in your blood. This blood will be analyzed i the laboratory at Virginia Commonwealth University and possibly at a future date at another institution. No names will be associated with the blood sample

ELIGIBILITY:
Inclusion Criteria:

* Men and Women over age of 18 non
* Women who are not pregnant
* Subject who are not prisoners
* Subjects presenting to the operation room for a Carotid artery stenting procedure
* Hemoglobin greater than or equal to 11mg/dl
* Subjects who speak english
* Subjects 18 years of age or older

Exclusion Criteria:

* Hemoglobin less than 11mg/dl
* Women who are pregnant
* Children under age of 18
* Prisoners
* Non English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for Carotid Stenting Procedure at Virginia Commonwealth University
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2011-03; Primary Completion 2013-10-09 (Actual); Study Completion 2013-10-09 (Actual)

PRIMARY OUTCOMES:
Biomarkers of Ischemia: Levels of Xanthine, Hypoxanthine and Inosine during Carotid Stenting Procedures | analysis will occur after all samples collected
  To compare a new blood test with can help the doctor determine if there is a brain injury or ischemia, The study will measure new biomarkers of neurologic stress called xanthine, hypoxanthine and inosine. Blood will be drawn as a part of the study to measure these biomarker levels in the blood. The blood will be analyzed in the laboratory at VCU.

CONTACTS AND LOCATIONS:
Overall Officials: Lynne Gehr, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States